CLINICAL TRIAL: NCT00609284
Title: Randomized Trial of Concomitant Chemotherapy in Patients With Locally Advanced HNSCC Treated by Radiotherapy-erbitux
Acronym: 2007-01
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Groupe Oncologie Radiotherapie Tete et Cou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GORTEC 2007-01
Record Dates: First submitted 2008-01-25; First posted 2008-02-07 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: HNSCC
Keywords: Stage III; Stage IV; locally advanced
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab; Carboplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Radiotherapy 70Gy, Erbitux, Carboplatin-5FU
  Interventions: Drug: cetuximab; Drug: Carboplatin, 5FU concomitant; Radiation: Radiotherapy
- 2 (Active Comparator): Radiotherapy 70Gy, Erbitux
  Interventions: Drug: cetuximab; Radiation: Radiotherapy

INTERVENTIONS:
Drug: cetuximab — D-7, D1, D8, D15, D22, D29, D43, D50
Drug: Carboplatin, 5FU concomitant — Carboplatin 70mg/m²/D ; 5FU 600 mg/m²/D, D1-4, D22-25, D43-46
  Arms: 1
Radiation: Radiotherapy — 70 Gy in 7 weeks

SUMMARY:
The aim of the trial is to study the efficacy of adding concomitant chemotherapy (carboplatin/5FU) to Erbitux-radiotherapy in patients with locally advanced head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* Squamous cell carcinoma of oral cavity, oropharynx, hypopharynx, larynx
* Stage III - IV (T0-T4, N0-N2b, M0)
* Not resected
* Karnofsky PS>=80
* Informed consent signed

Exclusion Criteria:

* Contra indication to chemotherapy or cetuximab

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2008-02-15 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 3 years

SECONDARY OUTCOMES:
Loco-regional control | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean BOURHIS, MD, PhD, Study Chair — GORTEC
Locations (5):
- France (5):
  - Centre hospitalier Annecy, Annecy
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Guillaume Le Conquerant, Le Havre
  - Centre hospitalier de Bretagne Sud, Lorient
  - Institut Gustave Roussy, Villejuif